CLINICAL TRIAL: NCT07095920
Title: Frequency-tuned Electromagnetic Field Treatment to Facilitate Recovery of Patients With Chronic Stroke
Brief Title: RESPARK - Brain Q for Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: BrainQ Technologies Ltd. (Industry); Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500526
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Chronic Stroke Patients; Cerebrovascular Accident (CVA)
Keywords: BrainQ; Electromagnetic Stimulation; upper extremity; rehabilitation; exercise; mobility
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BQ3.0 Active Stimulation (Experimental): 60 sessions over a period of 12 weeks (5 treatments per week) of active study intervention with the BQ 3.0 (frequency and intensity parameters will be set to 1-100 Hz.; 0.1-1.0 G), including a standardized, pre-defined and evidence-based physical and occupational therapy regimen concurrent with the study intervention.
  Interventions: Device: Device: Q Therapeutic System (BQ 3.0) - Active

INTERVENTIONS:
Device: Device: Q Therapeutic System (BQ 3.0) - Active — The BQ 3.0 is a medical device that produces and delivers non-invasive, extremely low intensity and frequency (1-100 Hz.; 0.1-1.0 G), frequency tuned electromagnetic fields in order to stimulate neuronal networks with the aim of reducing disability and promoting neurorecovery.

SUMMARY:
This trial tests a promising new intervention to promote post-stroke neural reorganization and functional recovery. The Q Therapeutic (BQ 3.0) is a wearable medical system that produces and delivers non-invasive, extremely-low-intensity and low-frequency, frequency-tuned electromagnetic fields in order to stimulate neuronal networks with the aim of reducing disability and promoting neurorecovery. This trial is a prospective, single-arm, open-label, single center clinical trial designed to evaluate the safety, feasibility, and efficacy of the Q Therapeutic (BQ 3.0) System in the rehabilitation of people with chronic stroke.

DETAILED DESCRIPTION:
The study intervention will consist of a total of 5 sessions per week over a period of 3 months (12 weeks) for a total of up to 60 sessions. Each participant must complete at least 40 sessions over the 12-week period to complete the protocol. No extra time will be given to complete all 60 sessions. Each session will last up to 60 minutes during which 40 minutes of active stimulation using the BQ 3.0 System will be administered to participants. The 40 minutes of stimulation will be paired with seated upper extremity (UE) exercises. Lastly, the device will be removed and 10 minutes of standing balance and LE strengthening exercises will be performed without stimulation. A battery of clinical assessments will be conducted before and after the 60 exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Upper Extremity Fugl-Meyer Assessment score between 22-50 (inclusive) of impaired limb.
2. Upper Extremity Fugl-Meyer Assessment score is within up to 3-point difference between Screening and Baseline visit.
3. Age 18 to 80 years of age (inclusive).
4. Stroke due to ischemia or to intracerebral hemorrhage.
5. >6 months to 5 years from stroke onset.
6. Box & Block Test score with affected arm is ≥1 block in 60 seconds.
7. Able to sit with the investigational system for 40 consecutive minutes.
8. Can follow a 3-step command, such as "take the paper, fold it in half, and return it to me", or a non-verbal equivalent.
9. Willingness to participate in physical exercises during study intervention sessions.
10. Availability of a relative or other caregiver that is able to participate in training and assist during treatment sessions at Brooks and home during the study duration.
11. If female, not pregnant or breastfeeding or planning pregnancy during the study period.
12. The subject is able to provide Informed consent.

Exclusion Criteria:

1. Severe neglect impairment interfering with assessments or treatments.
2. Severe depression, defined as Geriatric Depression Scale (GDS) Score >10/15
3. Presence of implanted or retained MR-incompatible devices or materials, or the presence of life-sustaining MR-compatible devices (e.g. pacemaker or internal cardiac defibrillator).
4. Active epilepsy or currently taking anti-epileptic medication (indicated for the treatment of a seizure disorder), or any epileptic seizure in the last 5 years
5. Botulinum toxin to the paretic arm: received in the prior 3 months OR expected before the 6-Month Visit
6. Severe upper extremity spasticity, defined as presence of contracture or modified Ashworth Scale score ≥3 in either biceps or pectoralis
7. Pre-existing neurological condition (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis, traumatic brain injury, spinal cord injury) or physical limitation that would interfere significantly with the subject's participation in the study and/or confound neurological or functional evaluation.
8. Significant visual disturbances, pre-existing or resulting from the index stroke, that cannot be corrected and that would interfere significantly with the subject's participation in the study and/or confound neurological or functional evaluation.
9. Unstable serious illness/condition (e.g., active cancer, severe heart failure, active major psychiatric condition) or life expectancy of less than 12 months.
10. Alcohol abuse and/or illicit drug abuse in the past 6 months, which is likely to influence ability to fully participate in the trial.
11. Participation in another trial that would conflict with the current study or clinical endpoint interference may occur.
12. Active participation in an upper extremity rehabilitation program provided by a licensed provider within 4 weeks from the screening visit and until the primary endpoint visit.
13. Employee of the Sponsor.
14. Prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment - Upper Extremity | Baseline, 3 months after, and 6 months after start of interventions
  A performance measure used to assess arm function. 33 items are scored on a scale of 0 to 2, where 0=cannot perform, 1=performs partially and 2=performs fully. An increase in score reflects an improvement in arm function.
Change from Baseline in Modified Rankin Scale (mRS) | Baseline, 3 months after, and 6 months after the start of interventions
  A 7-point scale used to measure the degree of disability or dependence in daily activities of people who have suffered a stroke. Scores range from 0 (no symptoms) to 6 (death). A decrease in score reflects a reduction in disability and improved independence.

SECONDARY OUTCOMES:
Cumulative incidence of adverse events | Initial consent through final study visit (6 months)
  The number of adverse events reported throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fox, PT, DPT, MHS, PhD, Principal Investigator — University of Florida & Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation Clinical Research Center, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with the study sponsor.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be shared from July 2025 to Dec 2026 between the site and study sponsor.
Access Criteria: De-identified data in excel spreadsheets will me made available to the study sponsor.